CLINICAL TRIAL: NCT07144644
Title: Surgical Efficiency and Postoperative Corneal Clarity With Near Physiologic vs High IOP Settings
Brief Title: 2311 TURGOR Study -Surgical Efficiency and Postoperative Corneal Clarity With Near Physiologic vs High IOP Settings
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2311
Record Dates: First submitted 2024-06-25; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-06

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Adjusting intraocular pressure (IOP) settings — Investigating whether adjusting IOP settings near physiologic levels during cataract surgery could potentially lead to better surgical outcomes

SUMMARY:
The study aims to investigate whether adjusting intraocular pressure (IOP) settings to near physiologic levels during cataract surgery could potentially lead to better surgical outcomes, particularly in terms of corneal clarity in the post-operative period.

DETAILED DESCRIPTION:
The study aims to investigate whether adjusting intraocular pressure (IOP) settings to near physiologic levels during cataract surgery could potentially lead to better surgical outcomes, particularly in terms of corneal clarity in the post-operative period. By comparing these two different IOP settings, we can determine the impact of IOP on surgical efficiency and the quality of post-operative results, especially in relation to corneal health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.
* Patients undergoing phacoemulsification surgery (OU) with or without femtosecond laser assistance (OU) with the Alcon Centurion system using Active Sentry handpieces (both eyes must undergo same treatment) . The cataract surgery and the use of the medical device(s) are planned by the principal investigator and are a part of regular care and are received regardless of being a part the study.
* Patients expected to undergo sequential cataract surgery in both eyes within 6 weeks of each other.
* Patients with the same LOCS III scale of nuclear portion of cataract in both eyes
* Patients whose eyes will both be operated by the same surgeon using a similar Centurion machine with similar wound architecture and size, viscoelastic, technique, and postoperative medications.
* Axial eye length cannot vary between eyes by more than 0.4 mm in an individual patient.
* At least 30% of patients with PanOptix, 30% Vivity and 30% monofocal IOLs (no mix and match)

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect the surgical outcome measures.
* Clinically significant ocular trauma.
* Patients with unusually dense cataract (4+ nuclear sclerosis), zonular instability, or pseudoexfoliation syndrome
* Patients requiring mechanical pupil expanding devices (iris hooks, Malyugin rings, etc.)
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL)
* Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure performed within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Reported pre-existing anxiety or pain disorder or history of psychiatric illness, chronic pain/narcotics, benzodiazepine usage.
* Epitheliopathy/ Epithelial complications intraoperatively that may in the opinion of the investigator affect corneal densitometry or edema postoperatively.
* Clinically significant IOL decentration
* Vulnerable populations which includes, but is not limited to potential subjects who are children, prisoners, pregnant women, mentally disabled persons, and economically and educationally disadvantaged persons.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This will be a multisite, prospective, randomized, contralateral-eye controlled, open-label clinical study, in which a maximum of 160 eyes will be treated with the Alcon Centurion System with Active Sentry during cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Central Corneal Thickness | 1 day following surgery for each eye
  Measurement by Pentacam

SECONDARY OUTCOMES:
Ocular Inflammation | 1 day following surgery for each eye
  Summed up inflammation score
Total BSS fluid usage during phaco emulsification | Day of surgery for each eye
  Balance salt solution fluid usage
Aspiration time | Day of surgery for each eye
  Aspiration Time

OTHER OUTCOMES:
BSS usage (Total) | Day of surgery for each eye
  Total BSS usage
Ultrasound time | Day of surgery for each eye
  Cumulative Dissipated Energy (CDE)
Use of opioids during cataract surgery | Day of surgery for each eye
  Opioid use
Incidence of reverse pupillary block during cataract surgery | Day of surgery for each eye
  Did this occur during surgery - yes or no
Uncorrected best corrected, and best corrected 25% low contrast visual acuity | At the 1 day postoperative, 7 days post operative, and 28 days post operative for each eye
  Best corrected vision
Grade of slit lamp corneal edema | 1 day following surgery for each eye
  Corneal edema grade
Corneal densitometry | At baseline, 1 day post-operative, and 7 day post-operative for each eye
  Corneal density
Change in the presence of posterior vitreous detachment/incidence | At baseline and 28 days post-operative of each eye
  Was there a change - yes or no

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Harvard Eye Associates
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States